CLINICAL TRIAL: NCT04354532
Title: Laparoscopic Banded Sleeve Gastrectomy: Single-Centre Experience With A 4-Year Follow-Up
Brief Title: Laparoscopic Banded Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Gentileschi, Head of Bariatric Unit, University of Rome Tor Vergata
Other Study IDs: UNRome
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Obesity, Morbid; Surgery
Keywords: Sleeve gastrectomy; Banded sleeve gastrectomy; Laparoscopy; Bariatric Surgery; Obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 209 patients were submitted to primary LBSG: All patients submitted to primary Laparoscopic Banded Sleeve Gastrectomy were examined. Collected data included demographic factors, pre-operative weight, pre-operative BMI, operative time, surgical complications, and clinical outcomes in terms of short and mid-term weight loss.
  Interventions: Procedure: Laparoscopic Banded Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Banded Sleeve Gastrectomy — The investigators performed Laparoscopic Sleeve Gastrectomy adding a MiniMizer Ring (Bariatric Solutions), a radiopaque silicone ring with four closing positions. The ring has a blue colour and for this reason it can easily be found back in revision surgery. The pulling lid is left in place with all closing positions in order to be adjusted postoperatively without having to place a new ring. The ring is slightly elastic and the fixation loops provide an anchorpoint to fix the ring in place which prevents it from slipping

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is now the most common bariatric procedure to treat morbidly obese patients. The main concern of LSG lies in the long-term weight regain which is reported to happen in up to 75.6% of patients after 6 years. The Investigators report the overall experience with Laparoscopic Banded Sleeve Gastrectomy (LBSG) using the Minimizer over a six-year period.

DETAILED DESCRIPTION:
Introduction. Laparoscopic sleeve gastrectomy (LSG) is now the most common bariatric procedure to treat morbidly obese patients. The main concern of LSG lies in the long-term weight regain which is reported to happen in up to 75.6% of patients after 6 years. The investigators report the overall experience with Laparoscopic Banded Sleeve Gastrectomy (LBSG) using the Minimizer over a six-year period.

Methods. The investigators performed a retrospective review of data from a prospectively collected database. All patients submitted to primary LBSG were examined. Patients were submitted to LBSG between February 2014 and January 2020. Collected data included demographic factors, pre-operative weight, pre-operative BMI, operative time, surgical complications, and clinical outcomes in terms of short and mid-term weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Severe Obesity with BMI > 35 kg/m2

Exclusion Criteria:

* Alcoholism
* Drug addiction
* Psychiatric Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients submitted to primary LBSG were examined. Patients were submitted to LBSG between February 2014 and January 2020. Collected data included demographic factors, pre-operative weight, pre-operative BMI, operative time, surgical complications, and clinical outcomes in terms of short and mid-term weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
% Excess Weight Loss | 4 years
  Weight loss after laparoscopic banded sleeve gastrectomy during the follow-up

SECONDARY OUTCOMES:
Post-operative complications | 4 years
  Complications occurred after laparoscopic banded sleeve gastrectomy during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: paolo gentileschi, MD, Principal Investigator — University Hospital of Tor Vergata, Rome, Italy
Locations (1):
- Michela Campanelli, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Welbourn R, Pournaras DJ, Dixon J, Higa K, Kinsman R, Ottosson J, Ramos A, van Wagensveld B, Walton P, Weiner R, Zundel N. Bariatric Surgery Worldwide: Baseline Demographic Description and One-Year Outcomes from the Second IFSO Global Registry Report 2013-2015. Obes Surg. 2018 Feb;28(2):313-322. doi: 10.1007/s11695-017-2845-9. PMID 28822052
- [Result] Lauti M, Kularatna M, Hill AG, MacCormick AD. Weight Regain Following Sleeve Gastrectomy-a Systematic Review. Obes Surg. 2016 Jun;26(6):1326-34. doi: 10.1007/s11695-016-2152-x. PMID 27048439
- [Result] Sarela AI, Dexter SP, O'Kane M, Menon A, McMahon MJ. Long-term follow-up after laparoscopic sleeve gastrectomy: 8-9-year results. Surg Obes Relat Dis. 2012 Nov-Dec;8(6):679-84. doi: 10.1016/j.soard.2011.06.020. Epub 2011 Jul 20. PMID 21890430
- [Result] Awad W, Garay A, Martinez C. Ten years experience of banded gastric bypass: does it make a difference? Obes Surg. 2012 Feb;22(2):271-8. doi: 10.1007/s11695-011-0555-2. PMID 22161231
- [Result] Lemmens L, Karcz WK, Bukhari W, Fink J, Kuesters S. Banded gastric bypass - four years follow up in a prospective multicenter analysis. BMC Surg. 2014 Nov 12;14:88. doi: 10.1186/1471-2482-14-88. PMID 25391401
- [Result] Fink JM, Hoffmann N, Kuesters S, Seifert G, Laessle C, Glatz T, Hopt UT, Konrad Karcz W, Marjanovic G. Banding the Sleeve Improves Weight Loss in Midterm Follow-up. Obes Surg. 2017 Apr;27(4):1098-1103. doi: 10.1007/s11695-017-2610-0. PMID 28214956
- [Result] Fink JM, von Pigenot A, Seifert G, Laessle C, Fichtner-Feigl S, Marjanovic G. Banded versus nonbanded sleeve gastrectomy: 5-year results of a matched-pair analysis. Surg Obes Relat Dis. 2019 Aug;15(8):1233-1238. doi: 10.1016/j.soard.2019.05.023. Epub 2019 May 24. PMID 31285129
- [Result] Parmar CD, Efeotor O, Ali A, Sufi P, Mahawar KK. Primary Banded Sleeve Gastrectomy: a Systematic Review. Obes Surg. 2019 Feb;29(2):698-704. doi: 10.1007/s11695-018-03626-1. PMID 30552547
- [Result] Tognoni V, Benavoli D, Bianciardi E, Perrone F, Ippoliti S, Gaspari A, Gentileschi P. Laparoscopic Sleeve Gastrectomy versus Laparoscopic Banded Sleeve Gastrectomy: First Prospective Pilot Randomized Study. Gastroenterol Res Pract. 2016;2016:6419603. doi: 10.1155/2016/6419603. Epub 2016 Apr 10. PMID 27143964
- [Result] Gentileschi P. Laparoscopic sleeve gastrectomy as a primary operation for morbid obesity: experience with 200 patients. Gastroenterol Res Pract. 2012;2012:801325. doi: 10.1155/2012/801325. Epub 2012 Jun 3. PMID 22701478
- [Result] Perrone F, Bianciardi E, Ippoliti S, Nardella J, Fabi F, Gentileschi P. Long-term effects of laparoscopic sleeve gastrectomy versus Roux-en-Y gastric bypass for the treatment of morbid obesity: a monocentric prospective study with minimum follow-up of 5 years. Updates Surg. 2017 Mar;69(1):101-107. doi: 10.1007/s13304-017-0426-z. Epub 2017 Mar 6. PMID 28266000
- [Result] Lemmens L, Van Den Bossche J, Zaveri H, Surve A. Banded Sleeve Gastrectomy: Better Long-Term Results? A Long-Term Cohort Study Until 5 Years Follow-Up in Obese and Superobese Patients. Obes Surg. 2018 Sep;28(9):2687-2695. doi: 10.1007/s11695-018-3248-2. PMID 29671124
- [Result] Filip S, Hutopila I, Copaescu C. Re-sleeve Gastrectomy - An Efficient Revisional Bariatric Procedure - 3 Years Results. Chirurgia (Bucur). 2019 Nov-Dec;114(6):809-823. doi: 10.21614/chirurgia.114.6.809. PMID 31928587
- [Result] Hanssen A, Plotnikov S, Acosta G, Nunez JT, Haddad J, Rodriguez C, Petrucci C, Hanssen D, Hanssen R. 3D Volumetry and its Correlation Between Postoperative Gastric Volume and Excess Weight Loss After Sleeve Gastrectomy. Obes Surg. 2018 Mar;28(3):775-780. doi: 10.1007/s11695-017-2927-8. PMID 28914408
- [Result] Cylke R, Skrzypek P, Ziemianski P, Domienik-Karlowicz J, Kosieradzki M, Lisik W. Single-anastomosis duodeno-ileal - new revision procedure in a patient with insufficient weight loss after sleeve gastrectomy. Wideochir Inne Tech Maloinwazyjne. 2018 Sep;13(3):407-411. doi: 10.5114/wiitm.2018.76686. Epub 2018 Jun 25. PMID 30302156
- [Result] Montuori M, Benavoli D, D'Ugo S, Di Benedetto L, Bianciardi E, Gaspari AL, Gentileschi P. Integrated Approaches for the Management of Staple Line Leaks following Sleeve Gastrectomy. J Obes. 2017;2017:4703236. doi: 10.1155/2017/4703236. Epub 2017 Feb 2. PMID 28261497
- [Result] Lemaitre F, Leger P, Nedelcu M, Nocca D. Laparoscopic sleeve gastrectomy in the South Pacific. Retrospective evaluation of 510 patients in a single institution. Int J Surg. 2016 Jun;30:1-6. doi: 10.1016/j.ijsu.2016.04.002. Epub 2016 Apr 8. PMID 27063637
- [Result] Gentileschi P, Kini S, Catarci M, Gagner M. Evidence-based medicine: open and laparoscopic bariatric surgery. Surg Endosc. 2002 May;16(5):736-44. doi: 10.1007/s00464-001-8239-y. Epub 2002 Jan 4. PMID 11997813
- [Derived] Gentileschi P, Benavoli D, Arcudi C, Campanelli M, Valente M, Petagna L, Bianciardi E. Laparoscopic Banded Sleeve Gastrectomy: Single-Center Experience with a Four-Year Follow-Up. J Laparoendosc Adv Surg Tech A. 2021 Nov;31(11):1269-1273. doi: 10.1089/lap.2020.0726. Epub 2021 Jan 15. PMID 33449836